CLINICAL TRIAL: NCT01345214
Title: An Open-label, Multiple-Dose Escalation Trial to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of ONO-7746 in Adult Cancer Patients With Chemotherapy Induced Thrombocytopenia
Brief Title: A Study of the Safety and Efficacy of ONO-7746 in Adult Cancer Patients With Chemotherapy Induced Thrombocytopenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to slow accrual of subjects.
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7746POU003
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Chemotherapy-Induced Thrombocytopenia
Keywords: ONO-7746; Chemotherapy Induced Thrombocytopenia; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E (Experimental)
  Interventions: Drug: ONO-7746

INTERVENTIONS:
Drug: ONO-7746 — 10mg, 20mg, 50mg, 100mg, 200mg and 300mg once-daily for 14 days

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ONO-7746 across multiple doses in patients with solid tumors and chemotherapy induced thrombocytopenia (CIT) scheduled to receive at least two cycles of myelosuppressive chemotherapy on Day 1 every 21 days at the same dosages and schedule in the study. The secondary objectives are to characterize the PK profiles of ONO-7746 and to explore the pharmacodynamic effect of ONO-7746 on CIT.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age ≥ 18 years
* Patients with confirmed solid tumor and scheduled to receive at least two cycles of myelosuppressive chemotherapy on Day 1 every 21 days at the same dosage and schedule in the study.
* Experienced thrombocytopenia as evidenced by a platelet count < 100 Gi/L in the preceding cycle immediately before study enrollment.
* ECOG performance status ≤ 2
* For females, surgically sterilized, postmenopausal or agree to use an acceptable form of birth control
* Patients treated with novel anticancer agents (e.g. bevacizumab, erlotinib, trastuzumab, cetuximab) may be allowed if it is considered the standard treatment by the investigator and after consultation and approval from the Sponsor
* PT/INR and aPTT are within 80% to 120% of the normal range

Exclusion Criteria:

* Experienced thrombocytopenia as evidenced by a platelet count < 25 Gi/L at any time in the preceding cycle immediately before enrollment into the study
* History or presence of clinically significant disease
* Received any TRAs, or rHuIL-11 within the last 4 weeks prior to screening
* Had received a bone marrow or peripheral blood stem cell infusion (within 1 year of screening).
* Pregnant, wanting to become pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-7746 across ascending multiple doses using vital signs, physical examinations, ECGs, ECOG performance status, CT/MRI, laboratory tests | up to four 21-day cycles (up to 84 days)

SECONDARY OUTCOMES:
Characterization of PK profiles on ONO-7746 and exploration of the PD effect of ONO-7746, including changes in platelet counts and any potential effects on ECGs | up to four 21-day cycles (up to 84 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (14):
- United States (3):
  - Fort Collins Clinical Site 13-01, Fort Collins, Colorado
  - Augusta Clinical Site 01-01, Augusta, Georgia
  - Ames Clinical Site 07-01, Ames, Iowa
- Russia (7):
  - Arkhangelsk Clinical Site 10-01, Arkhangelsk
  - Moscow Clinical Site 14-01, Moscow
  - St. Petersburg Clinical Site 11-01, Saint Petersburg
  - Samara Clinical Site 15-01, Samara
  - Tambov Clinical Site 16-01, Tambov
  - Tula Clinical Site 12-01, Tula
  - Ufa Clinical Site 17-01, Ufa
- South Korea (4):
  - Deagu Clinical Site 18-01, Deagu
  - Jeollanam-do Clinical Site 19-01, Jeollanam-do
  - Seoul Clinical Site 20-01, Seoul
  - Seoul Clinical Site 21-01, Seoul